CLINICAL TRIAL: NCT07368686
Title: A Prospective Clinical Study Evaluating the Effects of a Topical Multivitamin Serum on Facial Skin Hydration and Biophysical Parameters Following Microneedling
Brief Title: Topical Multivitamin Serum for Skin Heath
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-2025-VAMP-01
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Aesthetic
Keywords: Skin Heath; Topical; PDRN; Microneedeling; Skin Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biweekly Microneedeling - Group 1 (Active Comparator): Participants randomized to Group 1 will undergo an initial microneedling session using a hyaluronic acid vehicle solution to prime the skin. Subsequently, participants will undergo three (3) additional microneedling sessions utilizing the VAMP™ Advanced Multivitamin Serum, administered on a biweekly basis (every two weeks). In total, participants will receive four (4) microneedling treatment sessions, followed by two (2) follow-up visits
  Interventions: Device: Microneedeling with topical application of VAMP(TM) ADVANCED Topical Multivitamin Serum
- Monthly Microneedeling - Group 2 (Active Comparator): Participants randomized to Group 2 will undergo an initial microneedling session using a hyaluronic acid vehicle solution to prime the skin. Subsequently, participants will undergo three (3) additional microneedling sessions utilizing the VAMP™ Advanced Multivitamin Serum, administered on a monthly basis (every four weeks). In total, participants will receive four (4) microneedling treatment sessions, followed by two (2) follow-up visits.
  Interventions: Device: Microneedeling with topical application of VAMP(TM) ADVANCED Topical Multivitamin Serum

INTERVENTIONS:
Device: Microneedeling with topical application of VAMP(TM) ADVANCED Topical Multivitamin Serum — VAMP™ Topical Multivitamin Serum is not indicated for use in pregnancy, lactation, or in individuals under the age of 22. Female participants of childbearing potential will be required to undergo urine pregnancy testing at baseline and prior to each treatment session. They will also be instructed to use an acceptable form of effective contraception for the duration of the study.

SUMMARY:
Skin boosters are injectable and topical treatments designed to improve dermal quality and restore skin health. These products typically include hyaluronic acid formulations, biostimulatory agents, platelet-rich plasma (PRP), growth factors, and polynucleotides. Their growing use in aesthetic medicine is supported by their diverse mechanisms of action and routes of administration.

One such category of interest includes polynucleotide-based therapies, most notably Polydeoxyribonucleotide (PDRN). Derived from the DNA of salmon or trout, PDRN exhibits dual regenerative and anti-inflammatory properties. Mechanistically, it promotes tissue repair by supplying nucleotides essential for DNA synthesis and activates adenosine A2A receptors, thereby enhancing angiogenesis and mitigating inflammation. Clinically, PDRN has been applied in aesthetic medicine for skin rejuvenation, where it improves elasticity, texture, and reduces fine lines, as well as in wound healing and scar remodeling, supporting its integration into advanced bioregenerative protocols.

Among such agents, VAMP™ ADVANCED Topical Multivitamin Serum is formulated to improve hydration, elasticity, and overall skin radiance through a proprietary blend of amino acids, vitamins, and peptides. While preliminary data suggest potential benefits, robust peer-reviewed clinical studies remain limited. This study seeks to evaluate the efficacy of topical application of VAMP™ ADVANCED Topical Multivitamin Serum following microneedling in skin rejuvenation.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to adequately understand the verbal explanations and the written participant information provided in local language and ability and willingness to give consent to participate in the study. Signed and dated informed consent to participate in the study.
2. Participant interested in improving skin quality.
3. Immune-competent adult 22 years of age and older.
4. Has intent to undergo treatment to improve appearance of the facial skin.
5. Willingness to comply with pre-visit instructions, including shaving of facial area (for male participants), to allow for consistent biometric and photographic evaluations.
6. If the participant is a female of childbearing potential, she agrees to use an acceptable form of effective birth control for the duration of the study and is willing to take a urine pregnancy test (UPT) at Baseline and prior to receiving any study treatment.

   Acceptable forms of effective birth control include:
   * Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical caps) with spermicidal foam/gel/film/ cream/suppository;
   * Bilateral tubal ligation;
   * Combined oral contraceptives (estrogens and progesterone), implanted or injectable contraceptives on a stable dose for at least 28 days prior to Day 1;
   * Hormonal or copper intra uterine device (IUD) inserted at least 28 days prior to Day 1;
   * Vasectomized partner (in monogamous relationship) for at least 3 months prior to screening;
   * Strict abstinence (at least one month prior to Baseline and agrees to continue for the duration of the study or use acceptable form of birth control).
7. Negative UPT for women of childbearing potential at the Baseline visit.
8. Stable lifestyle and skincare regimen for at least 4 weeks

Exclusion Criteria:

1. Known or suspected allergy or hypersensitivity to any components of VAMP™ ADVANCED Topical Multivitamin Serum, including sodium hyaluronate, peptides, polynucleotides (e.g., PDRN), or excipients.
2. Known allergy or intolerance to topical anesthetics or lidocaine.
3. History of hypersensitivity reactions such as anaphylaxis, angioedema, or other severe allergic responses.
4. History of hypertrophic scarring, keloid formation, or post-inflammatory hyperpigmentation following cosmetic treatments.
5. Tattoos, piercings, or skin bleaching agents in the treatment area that may interfere with assessments, as judged by the Investigator.
6. Participants with known pigmentary instability or history of adverse response to microneedling.
7. Previous cosmetic or dermatologic procedures in the treatment area within the following time frames:
8. Previous treatment with cross-linked hyaluronic acid dermal fillers in the treatment area within the last 12 months.
9. Energy-based devices (laser, IPL, RF, ultrasound) in the last 6 months.
10. Microneedling, dermabrasion, mesotherapy, or chemical peels in the last 6 months.
11. Use of topical corticosteroids, retinoids, or depigmenting agents in the treatment area within the past 4 weeks.
12. Current use of immunosuppressive therapy, systemic corticosteroids, or chemotherapy within the last 3 months.
13. History of systemic autoimmune, collagen vascular, or bleeding disorders (e.g., lupus, scleroderma, thrombocytopenia).
14. Current pregnancy, positive urine pregnancy test at screening, breastfeeding, or intent to become pregnant during the study.
15. Participation in another clinical study within the past 30 days or concurrent participation in another interventional trial.
16. Any condition, including psychological, cognitive, or behavioral concerns, that would interfere with the ability to give informed consent, follow the protocol, or comply with follow-up requirements.
17. Initiation of a weight loss program or GLP-1 agonist therapy within 30 days before baseline or planned during study period.
18. Active skin conditions exacerbated by microneedling or transepidermal delivery, including chronic dermatitis or impaired barrier function.
19. Current participation by study personnel, immediate family members, or employees of the Sponsor.
20. Known allergy to fish or seafood, including but not limited to salmon, due to the potential presence of PDRN derived from marine sources.
21. History of cancer or previous radiation near or on the area to be treated.
22. Heavy smokers, classified as smoking more than 12 cigarettes per day.
23. Presence of any disease or lesions near or on the area to be treated, e.g.

    1. Inflammation, active or chronic infection in or near the treatment area
    2. Psoriasis, eczema, herpes zoster and acanthosis
    3. Cancer or precancerous condition (e.g. actinic keratosis)
    4. Severe skin laxity, flaccidity, or sagging
    5. Advanced photoaged/ photodamaged skin (e.g., advanced skin elastosis, multiple lentigo solaris lesions) or skin condition (e.g., very crinkled, very thin, fragile skin or severe skin atrophy) in the treatment area that in the Investigator's opinion could interfere with the safety or effectiveness of the study product or injection procedure.
24. Skin coloring/bleaching/tattoo in the treatment area, which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessment.
25. An underlying known disease, a surgical or medical condition that would expose the participant to undue risk, e.g. history of bleeding disorders, active hepatitis, active autoimmune disease such as connective tissue diseases, systemic lupus erythematosus, polymyositis, dermatomyositis, multiple sclerosis or scleroderma.
26. Use of concomitant medication that have the potential to prolong bleeding times such as anticoagulants or inhibitors of platelet aggregation (e.g., warfarin, clopidogrel, aspirin, baby aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), Omega 3 or Vitamin E), within 14 days prior to injection. Omega 3 and Vitamin E are acceptable only as part of a standard Topical Multivitamin formulation. Cyclooxygenase-2 (COX 2) inhibitors are allowed.
27. Treatment with chemotherapy, immunosuppressive agents, systemic corticosteroids within 3 months before treatment (inhaled or ophthalmic corticosteroids are allowed).
28. Use of hormonal therapy (ex. HRT or contraceptives) unless the participant has been on a stable dose for at least 3 months prior to screening and does not plan to make any changes to the HRT regimen during the study period.
29. Use of topical corticosteroids, topical prescription retinoids in the treatment area within 1 month of the Baseline visit or systemic retinoid treatment within 6 months of the baseline visit, or plan to receive such treatment.
30. Pregnancy (confirmed by positive urine pregnancy test (UPT)/ serum pregnancy test), breast feeding or intends to become pregnant over the duration of the study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Skin Hydration | Baseline to Week 10 (Group 1) and Week 16 (Group 2)
  The percentage change in skin hydration from baseline to Visit 6 will be assessed to compare the effects of biweekly versus monthly administration of VAMP™ Advanced following microneedling treatment. Assessment will be made using the Corneometer CM 825 (Courage+Khazaka electronic GmbH).

SECONDARY OUTCOMES:
Safety and Tolerability of Treatment | Baseline to Week 10 (Group 1) and Week 16 (Group 2)
  Incidence and frequency of adverse events
Global Aesthetic Improvement Scale (GAIS) Score Assessed by Blinded Evaluator | Baseline to Week 10 (Group 1) and Week 16 (Group 2)
  Proportion of participants rated as "improved" (improved, much improved, or very much improved) on the GAIS by a blinded evaluator at the end of the study
Participant Satisfaction With Treatment | Week 2 to Week 10 (Group 1) and from Week 4 to Week 16 (Group 2)
  Proportion of participants who report being at least "satisfied" (satisfied, very much satisfied, or extremely satisfied) on a seven-point participant satisfaction scale
Change in Transepidermal Water Loss (TEWL) From Baseline | Baseline to Week 10 (Group 1) and Week 16 (Group 2)
  Percentage change in TEWL from Baseline, measured using the Tewameter TM 21
Change in Skin Surface Biophysical Parameters From Baseline | Baseline to Week 10 (Group 1) and Week 16 (Group 2)
  Percentage change in surface evaluation of living skin cells (SELS: roughness, scaliness, smoothness, desquamation, and pore size), measured via the VisioScan VC 98.
Change in Skin Elasticity From Baseline | Baseline to Week 10 (Group 1) and Week 16 (Group 2)
  Percentage change in skin elasticity from Baseline, measured using the Cutometer Dual MPA 580.
Change in VISIA® CR Facial Imaging Metrics | Baseline to Week 10 (Group 1) and Week 16 (Group 2)
  Percentage change from Baseline in VISIA® CR-derived facial metrics as assessed by non invasive analysis of facial images

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, PhD, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No